CLINICAL TRIAL: NCT01685489
Title: A Phase 1b Dose Escalation Trial of PSK®/Placebo With Docetaxel to Treat Metastatic Castration-resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: funding sequestered
Sponsor: Bastyr University (Other)
Collaborators: University of Washington (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1U19AT006028-01A1 (NIH)
Record Dates: First submitted 2012-09-06; First posted 2012-09-14 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate; Neoplasm; Adenocarcinoma; Cancer; Metastatic; Castrate resistant; Docetaxel; PSK; Krestin; Trametes versicolor; Safety; Maximum tolerated dose; Mushroom; Natural; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Docetaxel; polysaccharide-K

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel, PSK® (Experimental): A 21-day lead-in oral PSK alone is followed by the addition of standard intravenous docetaxel at 75 mg/m2 evey 3 weeks for three cycles. After the third dose of docetaxel, study drug will be discontinued on day 14 to allow for a 7-day washout period before a fourth dose of docetaxel is administered.
  Interventions: Drug: Docetaxel, PSK®
- Docetaxel, Placebo (Placebo Comparator): A 21-day lead-in oral placebo alone is followed by the addition of standard intravenous docetaxel at 75 mg/m2 every 3 weeks for three cycles. After the third dose of docetaxel, the placebo will be discontinued on day 14 to allow for a 7-day washout period before a fourth dose of docetaxel is administered.
  Interventions: Drug: Docetaxel, Placebo

INTERVENTIONS:
Drug: Docetaxel, PSK®
  Other Names: Polysaccharide-K; Krestin; Polysaccharide-Kureha
  Arms: Docetaxel, PSK®
Drug: Docetaxel, Placebo
  Arms: Docetaxel, Placebo

SUMMARY:
This is a phase 1b study that follows a 3+3 dose escalation design and consists of a 21-day lead-in period of oral Polysaccharide Krestin (PSK)/placebo (study drug) alone followed by the addition to study drug of standard intravenous docetaxel at 75 mg/m2 every 3 weeks for three cycles. Study drug will be discontinued on day 15 of the third docetaxel cycle to allow for a 7-day washout period before the fourth dose of docetaxel. Pharmacokinetic (PK) analysis of docetaxel will be conducted during docetaxel cycle 1 (combination therapy) and cycle 4 (docetaxel alone). Serum for future PSK PK analysis will be collected on days 1, 3, and 15 of PSK/placebo lead-in and during cycles 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years or older
* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Evidence of metastatic disease by standard imaging studies (bone scan, Computerized Tomography Scan (CT) or Magnetic Resonance Imaging (MRI))
* Testosterone levels <50 ng/dL
* Confirmed progressive disease defined by one or more of the following:

  * an increase in PSA, > 2ng/dL x 2 or more values at least 1 week apart in the setting of metastatic disease
  * appearance of new bone lesions on bone scan
  * progression of soft tissue lesion defined by the Response Evaluation Criteria In Solid Tumors [RECIST] 1.1 criteria
* Concurrent use of an agent for testosterone suppression (e.g., Luteinizing Hormone Releasing Hormone [LHRH] agonist) if the patient is not surgically castrate
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 determined within 28 days before enrollment
* Recovery to CTCAE grade ≤ 1 toxicity, to patient's baseline status (except alopecia), or toxicities deemed irreversible from the effects of prior cancer therapy (CTCAEs grade > 1 that are not considered a safety risk by the investigator will be allowed)
* Adequate bone marrow function defined as:

  * absolute neutrophil count (ANC) > 1500 cells/mm³ without growth factor support
  * platelet count > 100,000 cells/mm³ without transfusion or growth factor support
  * hemoglobin > 9g/dL without transfusion or growth factor support
* Adequate liver function defined as:

  * total bilirubin < upper limit of normal (ULN)
  * alanine aminotransferase (ALT) < 1.5 x ULN
  * aspartate aminotransferase (AST) < 1.5 x ULN
* Adequate renal function defined as serum creatinine level within normal limits (WNL)
* At least a 6-month or greater life expectancy
* Ability to understand and sign a written informed consent, which will be obtained from study participants before undergoing any study-specific procedures
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
* Suitable venous access for the study-required blood sampling (i.e., including PK sampling)

Exclusion Criteria:

* Prior treatment with antineoplastic chemotherapy or radioisotopes for metastatic disease
* Prior adjuvant or neo-adjuvant chemotherapy within 12 months of study entry
* Last dose of sipuleucel-T therapy within 4 weeks of enrollment
* Any investigational therapies within 4 weeks of study entry
* Radiotherapy within 4 weeks of study entry
* Major surgery within 4 weeks of study entry, and not fully recovered to baseline or a stable clinical status
* Uncontrolled high blood pressure (systolic blood pressure > 160mmHg, diastolic blood pressure > 95mmHg)
* Receiving chronic steroid therapy. Topical and inhaled steroids are permitted
* Known severe hypersensitivity reactions to docetaxel or other drugs formulated in polysorbate 80, or to mushroom products
* Any comorbid condition or unresolved toxicity that would preclude administration of docetaxel
* Medical contraindication to any docetaxel pre-medications
* History of > grade 2 neurotoxicity or any toxicity from any cause that has not resolved to < grade 1
* Brain or other CNS metastasis
* The need for chronic daily immunosuppressive therapy, including concurrent use of prednisone
* Evidence of active second malignancy, except non-melanoma skin cancer
* Infection requiring intravenous antibiotic therapy or other severe infection within 14 days preceding first dose of study drug
* Inability to swallow oral medication or maintain a fast, as required 2 hours before and 1 hour after PSK administration
* Uncontrolled pain at baseline, impending complication from bone metastasis and/or presence of urinary obstruction
* Other medical or psychiatric condition that may increase the risk associated with trial participation or any other condition in the judgment of the investigator that may interfere with the interpretation of trial results or would make the patient inappropriate for enrollment in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05

PRIMARY OUTCOMES:
Determine tolerability dose of PSK alone and in combination with docetaxel | 42 days
  Adverse events are graded to determine a dose limiting toxicity of PSK during the lead-in PSK alone and during the docetaxel treatment in combination with PSK.
Determine maximum tolerated dose and recommended phase 2 dose of PSK in combination with docetaxel | 106 days
  When the maximum tolerated dose is determined, a total of 15 patients will be treated with the recommended phase 2 dose with the combination of docetaxel chemotherapy.

SECONDARY OUTCOMES:
Pharmacokinetics of docetaxel when combined with oral PSK | 106 days
  The plasma docetaxel levels are analyzed at eight time points during the cycle 1 of standard intravenous docetaxel at 75 mg/m2 with oral PSK/Placebo. After the seven-day washout of PSK/placebo at the cycle 3, the plasma docetaxel levels are analyzed again at eight time points during the cycle 4 of docetaxel treatment without PSK/Placebo.
Pharmacokinetics of oral PSK dosing and in combination with docetaxel | 106 days
  The serum PSK levels are analyzed at two time points during the lead-in cycle and eight time points during the cycle 1 of standard intravenous docetaxel at 75 mg/m2 with oral PSK/Placebo. After the seven-day washout of PSK/placebo at the cycle 3, the plasma docetaxel levels are analyzed again at eight time points during the cycle 4 of docetaxel treatment without PSK/Placebo.
Immunological laboratory analysis | 106 days
  Natural Killer (NK) cell functional activity, distributions of NK, B, and T cells, and IFN-gamma and TNF-alpha production capacity are analyzed and compared to those of the placebo group.
Clinical tumor markers | 106 days
  Circulating tumor cell (CTC) and prostate specific antigen (PSA) levels are compared to that of the placebo group during the oral PSK lead-in period and during the combination therapy with docetaxel and PSK.
Prostatic acid phosphatase | 106
  The serum level of prostatic acid phosphatase levels are compared to that of the placebo group during the oral PSK lead-in period and during the combination therapy with docetaxel and PSK.

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, MD, Study Director — Seattle Cancer Care Alliance - University of Washington; Cynthia A Wenner, Ph.D, Study Director — Bastyr University; Leanna J Standish, PhD, ND, LAc, Principal Investigator — Bastyr University; Mary (Nora) L Disis, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

REFERENCES:
- [Background] Antonarakis ES, Drake CG. Current status of immunological therapies for prostate cancer. Curr Opin Urol. 2010 May;20(3):241-6. doi: 10.1097/MOU.0b013e3283381793. PMID 20179598
- [Background] de Bono JS, Scher HI, Montgomery RB, Parker C, Miller MC, Tissing H, Doyle GV, Terstappen LW, Pienta KJ, Raghavan D. Circulating tumor cells predict survival benefit from treatment in metastatic castration-resistant prostate cancer. Clin Cancer Res. 2008 Oct 1;14(19):6302-9. doi: 10.1158/1078-0432.CCR-08-0872. PMID 18829513
- [Background] Fisher M, Yang LX. Anticancer effects and mechanisms of polysaccharide-K (PSK): implications of cancer immunotherapy. Anticancer Res. 2002 May-Jun;22(3):1737-54. PMID 12168863
- [Background] Fizazi K, Sternberg CN, Fitzpatrick JM, Watson RW, Tabesh M. Role of targeted therapy in the treatment of advanced prostate cancer. BJU Int. 2010 Mar;105(6):748-67. doi: 10.1111/j.1464-410X.2010.09236.x. PMID 20353536
- [Background] Fujita H, Ogawa K, Ikuzawa M, Muto S, Matsuki M, Nakajima S, Shimamura M, Togawa M, Yoshikumi C, Kawai Y. Effect of PSK, a protein-bound polysaccharide from Coriolus versicolor, on drug-metabolizing enzymes in sarcoma-180 bearing and normal mice. Int J Immunopharmacol. 1988;10(4):445-50. doi: 10.1016/0192-0561(88)90132-4. PMID 3139576
- [Background] Hurria A, Fleming MT, Baker SD, Kelly WK, Cutchall K, Panageas K, Caravelli J, Yeung H, Kris MG, Gomez J, Miller VA, D'Andrea G, Scher HI, Norton L, Hudis C. Pharmacokinetics and toxicity of weekly docetaxel in older patients. Clin Cancer Res. 2006 Oct 15;12(20 Pt 1):6100-5. doi: 10.1158/1078-0432.CCR-06-0200. PMID 17062686
- [Background] Iino Y, Yokoe T, Maemura M, Horiguchi J, Takei H, Ohwada S, Morishita Y. Immunochemotherapies versus chemotherapy as adjuvant treatment after curative resection of operable breast cancer. Anticancer Res. 1995 Nov-Dec;15(6B):2907-11. PMID 8669887
- [Background] Ikuzawa M, Matsunaga K, Nishiyama S, Nakajima S, Kobayashi Y, Andoh T, Kobayashi A, Ohhara M, Ohmura Y, Wada T, et al. Fate and distribution of an antitumor protein-bound polysaccharide PSK (Krestin). Int J Immunopharmacol. 1988;10(4):415-23. doi: 10.1016/0192-0561(88)90128-2. PMID 3170055
- [Background] Lu H, Yang Y, Gad E, Inatsuka C, Wenner CA, Disis ML, Standish LJ. TLR2 agonist PSK activates human NK cells and enhances the antitumor effect of HER2-targeted monoclonal antibody therapy. Clin Cancer Res. 2011 Nov 1;17(21):6742-53. doi: 10.1158/1078-0432.CCR-11-1142. Epub 2011 Sep 14. PMID 21918170
- [Background] Makkouk A, Abdelnoor AM. The potential use of Toll-like receptor (TLR) agonists and antagonists as prophylactic and/or therapeutic agents. Immunopharmacol Immunotoxicol. 2009;31(3):331-8. doi: 10.1080/08923970902802926. PMID 19555209
- [Background] Mickey DD, Bencuya PS, Foulkes K. Effects of the immunomodulator PSK on growth of human prostate adenocarcinoma in immunodeficient mice. Int J Immunopharmacol. 1989;11(7):829-38. doi: 10.1016/0192-0561(89)90137-9. PMID 2599718
- [Background] Nakazato H, Koike A, Saji S, Ogawa N, Sakamoto J. Efficacy of immunochemotherapy as adjuvant treatment after curative resection of gastric cancer. Study Group of Immunochemotherapy with PSK for Gastric Cancer. Lancet. 1994 May 7;343(8906):1122-6. doi: 10.1016/s0140-6736(94)90233-x. PMID 7910230
- [Background] Oba K, Teramukai S, Kobayashi M, Matsui T, Kodera Y, Sakamoto J. Efficacy of adjuvant immunochemotherapy with polysaccharide K for patients with curative resections of gastric cancer. Cancer Immunol Immunother. 2007 Jun;56(6):905-11. doi: 10.1007/s00262-006-0248-1. Epub 2006 Nov 15. PMID 17106715
- [Background] Odabasi Z, Mattiuzzi G, Estey E, Kantarjian H, Saeki F, Ridge RJ, Ketchum PA, Finkelman MA, Rex JH, Ostrosky-Zeichner L. Beta-D-glucan as a diagnostic adjunct for invasive fungal infections: validation, cutoff development, and performance in patients with acute myelogenous leukemia and myelodysplastic syndrome. Clin Infect Dis. 2004 Jul 15;39(2):199-205. doi: 10.1086/421944. Epub 2004 Jun 28. PMID 15307029
- [Background] Ostrosky-Zeichner L, Alexander BD, Kett DH, Vazquez J, Pappas PG, Saeki F, Ketchum PA, Wingard J, Schiff R, Tamura H, Finkelman MA, Rex JH. Multicenter clinical evaluation of the (1-->3) beta-D-glucan assay as an aid to diagnosis of fungal infections in humans. Clin Infect Dis. 2005 Sep 1;41(5):654-9. doi: 10.1086/432470. Epub 2005 Jul 21. PMID 16080087
- [Background] Sakamoto J, Morita S, Oba K, Matsui T, Kobayashi M, Nakazato H, Ohashi Y; Meta-Analysis Group of the Japanese Society for Cancer of the Colon Rectum. Efficacy of adjuvant immunochemotherapy with polysaccharide K for patients with curatively resected colorectal cancer: a meta-analysis of centrally randomized controlled clinical trials. Cancer Immunol Immunother. 2006 Apr;55(4):404-11. doi: 10.1007/s00262-005-0054-1. Epub 2005 Aug 20. PMID 16133112
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] van Zuylen L, Verweij J, Nooter K, Brouwer E, Stoter G, Sparreboom A. Role of intestinal P-glycoprotein in the plasma and fecal disposition of docetaxel in humans. Clin Cancer Res. 2000 Jul;6(7):2598-603. PMID 10914699
- [Background] Wenner CA, Martzen MR, Lu H, Verneris MR, Wang H, Slaton JW. Polysaccharide-K augments docetaxel-induced tumor suppression and antitumor immune response in an immunocompetent murine model of human prostate cancer. Int J Oncol. 2012 Apr;40(4):905-13. doi: 10.3892/ijo.2011.1292. Epub 2011 Dec 12. PMID 22159900
- [Background] Wils P, Phung-Ba V, Warnery A, Lechardeur D, Raeissi S, Hidalgo IJ, Scherman D. Polarized transport of docetaxel and vinblastine mediated by P-glycoprotein in human intestinal epithelial cell monolayers. Biochem Pharmacol. 1994 Oct 7;48(7):1528-30. doi: 10.1016/0006-2952(94)90580-0. PMID 7945455
- [Background] Zhou SF. Structure, function and regulation of P-glycoprotein and its clinical relevance in drug disposition. Xenobiotica. 2008 Jul;38(7-8):802-32. doi: 10.1080/00498250701867889. PMID 18668431
- See also: General information of Bastyr University — http://www.bastyr.edu